CLINICAL TRIAL: NCT03735030
Title: Comparative Bioavailability Study of Choriomon® (IBSA) Versus a Marketed hCG Formulation, Following Subcutaneous Administration in Healthy Women. Single-dose, Open-label, Randomized, Two-period, Two-way Cross-over, Bioavailability Study
Brief Title: Comparative Bioavailability Study of Human Chorionic Gonadotropin (hCG)-IBSA Versus a Marketed hCG Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18CH-hCG09
Record Dates: First submitted 2018-10-31; First posted 2018-11-08 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- human hCG (Experimental)
  Interventions: Drug: Human hCG 10'000 IU
- recombinant hCG (Active Comparator)
  Interventions: Drug: Recombinant hCG 6'500 IU

INTERVENTIONS:
Drug: Human hCG 10'000 IU — A single dose of 10'000 IU of human hCG will be injected in 24 healthy subject volunteers.
  Arms: human hCG
Drug: Recombinant hCG 6'500 IU — A single dose of 6'500 IU recombinant hCG will be injected in 24 healthy subject volunteers.
  Arms: recombinant hCG

SUMMARY:
In the present study, the rate and extent of hCG absorption will be compared between the two treatments in healthy women aged 20 to 45 years.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the study;
2. Sex and Age: healthy pre-menopausal women, 20-45 years old inclusive;
3. Body Mass Index: 18.5-30 kg/m2 inclusive;
4. Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, heart rate 50-90 bpm, measured after 5 min at rest in the sitting position;
5. Hormonal oral contraceptives: Combined oral contraceptive pill for at least 2 months before the screening visit;
6. Menstrual cycle: history of a normal menstrual cycle before combined oral contraceptive pill use;
7. hCG: endogenous hCG levels <1.2 IU/L at screening and Day -1, Period 1;
8. Pituitary down-regulation: Luteinizing hormone (LH) <5 IU/L; Follicle stimulating hormone (FSH) <4 IU/L at Day -1, Period 1;
9. Papanicolaou smear (PAP) test: negative or not clinically significant PAP test results within 12 months before the screening visit or at screening;
10. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study;
11. Additional contraception: study participants with an active sexual life must be using one additional contraceptive method, as follows:

    1. A male sexual partner who agrees to use a male condom with spermicide
    2. A sterile sexual partner.

Exclusion Criteria:

1. Contraindications: any contraindications to combined oral contraceptive pill or gonadotropins;
2. Electrocardiogram 12-leads (supine position): clinically significant abnormalities;
3. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study;
4. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness;
5. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study;
6. Diseases: relevant history of cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, immunological, dermatological, endocrine, genitourinary (e.g. polycystic ovary disease, ovarian cysts, primary ovarian failure, early menopause or abnormal bleeding of undetermined origin), malignant neoplasia, neurological or psychiatric diseases that could interfere with the aim of the study;
7. Medications: treatment with gonadotropin preparations within 6 months prior to screening; other medications, including over the counter medications and herbal remedies, for 2 weeks before the start of the study;
8. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study;
9. Blood donation: blood donations for 3 months before this study;
10. Drug, alcohol, caffeine, tobacco: history of drug, alcohol (>1 drink/day defined according to the United Stated Department of Agriculture (USDA) Dietary Guidelines 2015-2020; 17), caffeine (>5 cups coffee/tea/day) or tobacco abuse (≥10 cigarettes/day);
11. Drug test: positive result at the drug test at screening or day -1, Period 1;
12. Alcohol test: positive alcohol breath test on day -1;
13. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians;
14. Pregnancy: positive or missing pregnancy test at screening or at day -1 of each period; pregnant or lactating women.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Rate of absorption (Cmax) | 192 hours post dose
  To assess the bioavailability of the test and reference products in terms of rate (baseline-corrected, dose-normalised Cmax) of hCG absorption after single s.c. injection to healthy female subjects.
Extent of absorption (AUC0-t), Area under the concentration-time curve | 192 hours post dose
  To assess the bioavailability of the test and reference products in terms of extent (baseline-corrected, dose-normalised AUC0-t) of hCG absorption after single s.c. injection to healthy female subjects.Area under the concentration-time curve from administration to the last observed concentration time t, calculated with the linear trapezoidal method.

SECONDARY OUTCOMES:
t1/2: Half-life | 192 hours post dose
  To evaluate the baseline-corrected, dose-normalised (when applicable) t1/2 (Half-life) value after single dose administration of test and reference products;
Tmax: Time to achieve Cmax | 192 hours post dose
  To evaluate the baseline-corrected, dose-normalised (when applicable) Tmax value after single dose administration of test and reference products;
AUC0-∞: Area under the concentration-time curve extrapolated to infinity | 192 hours post dose
Frel : Relative bioavailability | 192 hours post dose
  calculated as dose-normalised ratio AUC0-t (T)/dose(T) / AUC0-t (R)/dose(R)
Treatment emergent adverse events (TEAEs) | through study completion up to 46 days.
  percentage of subjects with any TEAE

CONTACTS AND LOCATIONS:
Locations (1):
- CROSS Research SA, Arzo, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Radicioni M, Leuratti C, Cometti B. Randomized Pharmacokinetic Study of a Highly Purified Human Chorionic Gonadotropin and of a Recombinant Human Chorionic Gonadotropin Following Single Subcutaneous Administration in Healthy Women. Clin Drug Investig. 2022 Mar;42(3):199-206. doi: 10.1007/s40261-022-01118-w. Epub 2022 Feb 9. PMID 35137345